CLINICAL TRIAL: NCT05406544
Title: Df-Life : Quality of Life in Patients With Fibrous Dysplasia
Acronym: Df-Life
Status: Completed | Type: Observational
Sponsor: Hospices Civils de Lyon (Other)
Responsible Party: Sponsor
Other Study IDs: 69HCL22_0374; 2022-A01239-34 (Other: ID RCB)
Record Dates: First submitted 2022-06-02; First posted 2022-06-06 (Actual); Last update posted 2024-03-22 (Actual); Status verified 2024-03

CONDITIONS: Fibrous Dysplasia
Keywords: Fibrous dysplasia; quality of life
MeSH Terms: conditions — Fibrous Dysplasia of Bone | interventions — Smell

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (3):
- FD qualitative study on quality of life.: FD patients (FD monostotic, FD polyostotic, with or without craniofacial damages) will be invited to attend a focus group on the following themes: symptoms, self-image, psychological and emotional well-being, difficulties in daily life and adaptative strategies. The focus-groups will be conducted in a semi-directive manner by a moderator and will be recorded; after a verbatim transcription of the focus group recordings, the data will be analyzed manually and with the help of a semantic analysis software. It will allow common notions about quality of life in FD to emerge. A demographic questionnaire will also be completed by the participants.
  Interventions: Other: FD qualitative study on quality of life
- FD quantitative sudy on quality of life and olfaction.: Participants will receive two questionnaires to complete: the SF36 questionnaire (quality of life) and the SELF-MOQ questionnaire (olfaction impairment evaluation). Other data required for the study will be extracted from the medical record: age, weight, height, affected bone sites, Radiological/ biological activity data, sensorial deficit, medication. A demographic questionnaire will also be completed.
  Interventions: Other: FD quantitative sudy on quality of life and olfaction.
- FD qualitative and quantitative study on quality of life and olfaction.: Patients will be invited to attend a focus group on quality of life (qualitative study) as described for group 1 and to complete questionnaires on quality of life and olfaction (quantitative study) as described for group 2
  Interventions: Other: FD qualitative study on quality of life; Other: FD quantitative sudy on quality of life and olfaction.

INTERVENTIONS:
Other: FD qualitative study on quality of life — Patients will be contacted and focus groups will be organized with 6 to 8 patients presenting different types of FD: monostotic, polyostotic, with or without craniofacial damage. Several focus-groups will be conducted with men only or women only. Patients will be led in a semi-directive manner by a moderator who will use an interview grid listing all the topics to be addressed: symptoms, self-image, psychological and emotional well-being, difficulties in daily life and adaptative strategies. The discussions will be recorded and transcribed verbatim. Data will be analyzed manually by 2 investigators and with the help of a semantic analysis software. The objective is to bring out common notions about the quality of life of patients, their psychological and emotional well-being, their difficulties in daily life and their coping strategies according to their condition. Differences or similarities between men and women will be investigated.
  Groups: FD qualitative and quantitative study on quality of life and olfaction.; FD qualitative study on quality of life.
Other: FD quantitative sudy on quality of life and olfaction. — Participants will receive 3 questionnaires to complete: the SF36 questionnaire (quality of life), the SELF-MOQ questionnaire (olfaction evaluation) and a demographic questionnaire. Other data required for the study will be extracted from the medical record: age, weight, height, affected bone sites, Radiological/ biological activity data, sensorial deficit, medication. For each questionnaire, scores will be calculated and compared between the different FD patient populations according to sex, age and type of FD.
  Groups: FD qualitative and quantitative study on quality of life and olfaction.; FD quantitative sudy on quality of life and olfaction.

SUMMARY:
Fibrous dysplasia (FD) is a congenital skeletal disorder with multiple complications such as bone pain, fractures, deformities and nerve compression. Few quantitative studies have demonstrated its physical, mental and social negative impacts on patients but none have qualitatively evaluated their global quality of life. Our hypothesis is that a better knowledge of the quality of life of FD patients should allow to target the actions to be implemented to improve patients'care.

The main objective of this qualitative research is therefore to investigate the quality of life of FD patients through 2 approaches: a qualitative study with focus groups interviews addressing several themes: self-image, psychological and emotional well-being, difficulties and adaptative strategies; and a quantitative study to measure the impact of FD on quality of life and on olfaction (sometimes affected by nerve compression due to the disease) using standardized questionnaires Short Form 36 (SF36) and Self-reported Mini Olfactory Questionnaire (SELF-MOQ).

ELIGIBILITY:
Inclusion Criteria:

* Men and women
* 18 years and more
* with Fibrous dysplasia
* Being followed in the rheumatology Department of the E. Herriot Hospital in Lyon.
* Non-opposition to take part in the study
* written consent to the audio recording of the discussions.

Exclusion Criteria:

* Legal incapacity or limited legal capacity
* Psychiatric or neurological condition that severely impairs comprehension
* Difficulty understanding spoken French
* Patients with another pathology with a major impact on quality of life

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Primary care clinics: adults coming for consultation or hospitalization for fibrous dysplasia in Hopital Edouard Herriot rheumatology department in Lyon, France.
Sampling Method: Non-Probability Sample
Enrollment: 149 (Actual)
Dates: Start 2022-11-28 (Actual); Primary Completion 2022-11-28 (Actual); Study Completion 2023-05-02 (Actual)

PRIMARY OUTCOMES:
FD Qualitative study: notions on quality of life | during group interview (90 minutes)
  quality of life concepts that will emerge during group interviews.
FD Quantitative study: scores of quality of life and olfaction impairment | during 30 minutes
  quality of life measured with SF36 score. Patients will answer to 11 questions. Olfaction impairment measured with SELF-MOQ olfaction score. Patients will answer to 14 questions

CONTACTS AND LOCATIONS:
Overall Officials: Roland CHAPURLAT, Pr, Principal Investigator — Hospices Civils de Lyon
Locations (1):
- Edouard Herriot Hospital - rheumatology, Lyon, France